CLINICAL TRIAL: NCT06827366
Title: Lifestyle Intervention Among Participants of the French Colorectal Cancer Screening Program (LIFE-SCREEN)
Acronym: LIFE-SCREEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: International Agency for Research on Cancer (Other); University of Bordeaux (Other); Hôpital Edouard Herriot (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIFE-SCREEN (ET 24-226)
Record Dates: First submitted 2024-10-24; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer Prevention; Colorectal Cancer
Keywords: colorectal cancer; primary prevention; screening; physical activity; nutrition; recommendations
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Colorectal cancer free participants receive the 'usual care' following a positive FIT test and diagnostic colonoscopy
- Intervention (Active Comparator): Colorectal cancer free participants receive evidence-based diet and lifestyle advice in addition to the 'usual care' following a positive FIT test and diagnostic colonoscopy
  Interventions: Behavioral: Diet and lifestyle advice following a positive FIT test and diagnostic colonoscopy

INTERVENTIONS:
Behavioral: Diet and lifestyle advice following a positive FIT test and diagnostic colonoscopy — Participants will be recruited during CRC screening and will be included if they have a positive faecal immunochemical test (FIT) and are diagnosed with adenomas but are CRC negative during the colonoscopy. Participants receive evidence-based diet and lifestyle advice intervention with 'usual care'
  Arms: Intervention

SUMMARY:
The investigators propose a randomized controlled trial to develop and evaluate the impact of promoting advice on diet and lifestyle recommendations for cancer prevention at colorectal cancer screening among individuals who may be at higher risk for colorectal cancer (CRC). The specific objectives of this study are to 1) develop a lifestyle intervention based on evidenced-based diet and lifestyle recommendations (i.e. those proposed by the World Cancer Research Fund (WCRF) and the French National Cancer Institute); 2) evaluate the effect of the intervention on the adherence to the target diet and lifestyle recommendations as well as other subjective health measures, including quality of life; 3) evaluate the effect of the intervention on anthropometrics.

DETAILED DESCRIPTION:
A pilot study was launched on March 23rd 2022 to assess the feasibility and acceptance of the LIFE-SCREEN study protocol. During the pilot study, participants were asked to complete several questionnaires about their lifestyle and health, while also having their anthropometrics measured and optional their blood taken and faecal sample collected. Evaluation questionnaires were completed by all participants and some participated in focus group meetings. Based upon this pilot study, it was decided in 2024 to drop the biospecimen collections due to feasibility issues.

This RCT study launched in November 2024 will be a parallel, two-arm, randomized controlled trial (RCT) in individuals at higher risk of colorectal cancer (CRC), comparing an evidence-based diet and lifestyle advice intervention with 'usual care'. Participants will be recruited during CRC screening and will be included if they have a positive faecal immunochemical test (FIT) and are diagnosed with adenomas but are CRC negative during the colonoscopy. The advice provided will be developed based on the World Cancer Research Fund (WCRF) & French National Cancer Institute (INCA) evidence-based diet and lifestyle recommendations using the habit-theory and will be delivered using multiple materials (e.g. leaflets, posters and digital information) by health professionals in hospitals based in the Rhone region, France. Invitation to participate in the trial will be performed by the gastroenterologist during the clinical visit to provide information on colonoscopy, but the delivery of the intervention and baseline measurement will happen two to three weeks after the colonoscopy. Data will be collected at baseline, 3, 6 and 12 months. At baseline, participants will be required to answer questionnaires on sociodemographic and medical history. At all aforementioned time points, online or paper-based questionnaires will be administered to collect information on diet and lifestyle behaviours, knowledge on healthy lifestyle, quality of life and medical therapy. Participants will also have their anthropometric measured during baseline and follow-up appointments. The primary outcome of this intervention will be adherence to target recommendations at 3 months and beyond. Univariate and multivariate statistical analyses as well as qualitative analyses will be performed.

Providing lifestyle advice for cancer prevention at screening programs is a new field in public health that has the potential to be cost-effective, convenient, appealing and widereaching. It may also help to reach individuals at higher risk at a time-window when they adherence to cancer prevention recommendations, as well as on quality of life and body weight among individuals at higher risk of CRC.

ELIGIBILITY:
Inclusion Criteria:

* Having read the information note and agreeing to participate
* Will and availability to be committed for a full year
* At high risk for CRC but CRC negative
* Affiliated to a health security system
* Having a score on the adherence to the recommendation lower than or equal to 7 out of 9 at baseline.
* Able to read, write and understand French

Exclusion Criteria:

* Under a strict diet such as meal replacements, diets for co-morbidities such as diabetes
* Immobile due to physical constraints (e.g. handicap that is not compatible with physical activities)
* Extensive intestinal surgery such as colectomy or surgical resection of the colon
* Chronic gastrointestinal illness (IBD, IBS, celiac disease)
* Colorectal cancer confirmed or history of a primary cancer
* Severe malnutrition
* Pregnant
* Participation in another lifestyle study

NB : For this study, there is no exclusion period from other research, and participants can simultaneously take part in another study unless it concerns lifestyle.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to the evidence-based lifestyle recommendations | 3 months
  The primary outcome of the trial will be adherence to the evidence-based lifestyle recommendations (expressed as an adherence score on the individual lifestyle recommendations).
  Score :
  * unabbreviated scale title : World Cancer Research Fund's (WCRF)
  * minimum value = 0 (more unhealthy behaviours) / maximum value = 7 (more healthy behaviours)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Huybretchts, PhD, Study Director — International Agency Research Cancer
Locations (1):
- Centre Léon Bérard, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No